CLINICAL TRIAL: NCT06382727
Title: CONTINUation of Enteral Nutrition Prior to Extubation Compared to Standard Care: a Pilot Randomised Controlled Trial (CONTINUE Trial)
Brief Title: CONTINUation of Enteral Nutrition Prior to Extubation Compared to Standard Care
Acronym: CONTINUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emma Ridley (Other)
Responsible Party: Sponsor-Investigator, Emma Ridley, A/Prof, The Alfred
Organization: The Alfred (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ANZIC- RC ER008
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Critical Illness
Keywords: Extubation; Enteral Nutrition; Fasting
MeSH Terms: conditions — Critical Illness; Fasting

STUDY DESIGN:
Intervention Model Description: CONTINUE is a multi-centre, open-label, prospective parallel, pilot randomised controlled trial being conducted in Australia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Continuation of enteral nutrition (EN) prior to extubation (Experimental): Maintenance of EN at the same hourly rate until the point of extubation. Maximal suction of the EN tube prior to extubation will take place.
  Interventions: Other: EN will be continued up to extubation (EN will not be withheld prior to extubation)
- Control group: Cessation of EN prior to extubation (No Intervention): Cessation of EN at least 4-6 hours prior to the point of extubation. Maximal suction of the EN tube prior to extubation will take place.

INTERVENTIONS:
Other: EN will be continued up to extubation (EN will not be withheld prior to extubation) — As per the arm/group descriptions.
  Arms: Intervention group: Continuation of enteral nutrition (EN) prior to extubation

SUMMARY:
Critically ill patients admitted to the Intensive Care Unit (ICU) often need to be connected to a breathing machine (ventilator) and are unable to eat. During this time, liquid nutrition is delivered via a feeding tube to the stomach or bowel (termed enteral nutrition (EN)) to ensure nutrition needs are provided until such time that the patient can eat normally.

The delivery of nutrition via EN is frequently interrupted due to procedures and changes in the gastrointestinal system that can cause digestion to be slow. One of the main contributors to EN interruptions is fasting prior to removal of the breathing tube (termed extubation).

The practice of pausing EN prior to the removal of the breathing tube is historical and based on evidence for patients who are not within the ICU. There is currently no scientific consensus on whether pausing of EN is necessary, or for how long. Because of this, some clinicians choose to pause EN prior to removal of the breathing tube and some clinicians continue to provide EN.

This study is a pilot randomised controlled trial of fasting patients for at least 4 hours prior to removal of the breathing tube compared with not pausing EN. The investigators hypothesise that this will reduce the number of hours of fasting in the 24 hours prior to extubation.

DETAILED DESCRIPTION:
The provision of EN is standard practice to mechanically ventilated patients within the ICU. Delivery is frequently interrupted, with patients often receiving approximately half of prescribed volumes. One of the main contributors to this is fasting prior to extubation. Fasting prior to extubation is historically informed from pre-anaesthetic practice in patients who are not critically ill where fasting allows for adequate gastric emptying and reduces the risk of aspiration on induction. The practice of fasting prior to extubation is less informed, and variable. A recent scoping review identified only 1 randomised controlled trial (RCT) and 13 observational studies on this topic. The review found fasting durations varied between 0-34 hours and the reasons for fasting prior to extubation were safety related; however, these reasons were often extrapolated from data outside of the ICU as outlined above. The review concluded that there is an evidence gap and no evidence-based consensus as to the rationale and duration of fasting critically ill patients prior to extubation.

The clinical consequences of fasting (and particularly repeated fasting) are not well understood; however, it is known that fasting leads to reduced nutrition which may negatively impact response to illness, particularly in patients with a long length of stay. Beyond this, the requirement for fasting may delay extubation and progression of care (as extubation may be cancelled if the patient is not adequately fasted) and lead to unnecessary use for nursing and medical resources.

The CONTINUE trial represents the first trial of its kind in Australia and seeks to determine feasibility to inform a program of research that addresses a universal practice for critically ill patients requiring mechanical ventilation. Establishment of feasibility will provide data to inform a large RCT of similar nature, powered to determine differences in important clinical outcomes such as reintubation rate, ventilator free days to day 28 of admission and development of aspiration pneumonia. The culmination of this research will be to create an evidence-based guideline on pre-extubation fasting with the aim of standardising and informing international practice.

The primary aim is to determine whether continuing EN to the point of extubation and performing maximal nasogastric aspiration immediately prior is feasible and decreases total fasting in the time 24 hours prior to extubation compared to standard practice of ceasing EN 4- 6 hours prior to planned extubation, in low risk ventilated patients. Secondary objectives include assessment of important safety related endpoints including change in oxygenation requirements, aspiration, reintubation rate at 48 hours after extubation and clinical outcome measures including ICU and hospital morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Receiving invasive mechanical ventilation > 24 hours and < 10 days in the index ICU admission
* Receiving EN at a rate ≥ 30ml/hr
* Planned for extubation within the hours of 0800-1800

Exclusion Criteria:

* EN delivery via a fine bore nasogastric tube that is unable to be aspirated
* A single gastric residual volume ≥ the maximum protocol limit at the participating site has been recorded within the last 24 hours
* Currently receiving extracorporeal membrane oxygenation
* Acute neurological pathology
* A time critical medication is required via the enteral route (including anti-parkinsons and immunosuppressant medication) and no adjustments can be made
* Pre-existing swallow, bulbar dysfunction and/or concern around inadequate airway protection
* A laparotomy has been performed within 72 hours of planned extubation
* Confirmed pregnancy
* Patient not deemed appropriate to be reintubated in the event of deterioration
* Treating clinician believes enrolment is not in the best interests of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Fasting time (hours) | 24 hours prior to endotracheal tube removal
  Fasting time due to planned extubation

SECONDARY OUTCOMES:
Reintubation rate | 48 hours post endotracheal tube removal
  Actual reintubation rate and according to an objective criterion for failure:
  Respiratory acidosis (pH <7.35 with Paco2 >45 mm Hg); Spo2 less than 90% or Pao2 less than 60 mm Hg at Fio2 greater than 0.4; Respiratory rate greater than 35/min; Decreased level of consciousness (defined as a decrease in GCS score >1 point); Agitation, or clinical signs suggestive of respiratory muscle fatigue, increased work of breathing (eg, the use of respiratory accessory muscles, paradoxical abdominal motion, or retraction of the intercostal spaces), or both; Patients dying within 72 hours will also be considered as extubation failures.
Days alive and free of mechanical ventilation | Up to day 28 post randomisation
  Number of days alive and free of mechanical ventilation
Commencement of antibiotics | Up to 7 days post endotracheal tube removal
  Commencement of antibiotics for a chest infection or aspiration
Ratio of oxygen saturation (SpO2)/ fraction of inspired oxygen (FiO2) | 12 hours post endotracheal tube removal
  SpO2:FiO2 ratio
ICU length of stay | Up to day 28 post randomisation
  ICU length of stay (days)
In-hospital mortality | Up to day 28 post randomisation
  In-hospital mortality during ICU or acute ward admission
Nutrition delivery | 24 hours prior to endotracheal tube removal
  The absolute and relative (to calculated requirements) amount of calories delivered
Recruitment rate | Up to the end of the study period
  Number of patients recruited per month
Protocol compliance | Up to Endotracheal Tube removal
  Defined as the proportion of patients receiving the allocated intervention

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Gold Coast University Hospital, Southport, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Varghese JA, Tatucu-Babet OA, Miller E, Lambell K, Deane AM, Burrell AJC, Ridley EJ. Fasting practices of enteral nutrition delivery for airway procedures in critically ill adult patients: A scoping review. J Crit Care. 2022 Dec;72:154144. doi: 10.1016/j.jcrc.2022.154144. Epub 2022 Sep 15. PMID 36115335